CLINICAL TRIAL: NCT02088814
Title: Prevention of Posttraumatic Stress Symptoms in Young Children With Burns: a Randomized Controlled Trial
Acronym: EPICAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Markus A. Landolt, Prof. Markus Landolt, PhD, University Children's Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 100014_149158
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Burns
Keywords: posttraumatic stress; burns; injuries; children
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'EPICAP' (Experimental): Secondary preventive psychological intervention with parents of children ages 1-4 with acute burn injuries, consisting of psychoeducation, trauma narrative, storybook, provision of coping skills
  Interventions: Behavioral: 'EPICAP'
- Medical treatment as usual (No Intervention): Medical treatment of burn injuries as usual

INTERVENTIONS:
Behavioral: 'EPICAP' — standardized, secondary preventive psychological intervention with parents of children ages 1-4 with acute burn injuries, consisting of psychoeducation, trauma narrative, storybook, provision of coping skills
  Arms: 'EPICAP'

SUMMARY:
Background: Previous studies have found considerable rates of posttraumatic stress disorder (PTSD) or clinically relevant posttraumatic stress symptoms (PTSS) in preschoolers with injuries following accidental trauma. In consequence, secondary preventive efforts (early interventions) should be undertaken to minimize such long-term deleterious consequences in children.

Aims: The proposed study aims at examining the effect of a newly developed, standardized early psychological intervention in reducing posttraumatic maladjustment and in enhancing health-related quality of life in children ages 1 to 4 years with acute burn injuries.

Method: The study is designed as a randomized controlled trial within a stepped procedure. First, eligible children will be screened 5 to 7 days post injury by means of a standardized measure for their risk of developing PTSS. After a baseline assessment, children at risk will then be randomly allocated to either a control group (standard medical care) or an intervention group. Participants of the intervention group will be provided with the standardized "EPICAP 1-4" intervention which uses established cognitive-behavioral techniques and is directed to the parents. The intervention consists of two face-to-face sessions (at baseline and 1 week later) and a follow-up call or short follow-up face-to-face meeting (6 weeks after the first session). Blinded follow- up assessments with standardized parent report measures will be conducted at 3 and 6 months post injury. The primary outcome measures are child PTSD and PTSS, secondary outcome measures include child behavior and health-related quality of life. In addition, a variety of socio-demographic, medical and parental variables will be assessed as co-variates. Children screened as low-risk will be reassessed only at 6 months to make sure that the screening procedure is valid.

DETAILED DESCRIPTION:
Background: Unintentional injuries in preschoolers are frequent. Many accidents meet criteria for a psychotraumatic event as defined by the DSM-IV. It is therefore not surprising that previous studies have found considerable rates of posttraumatic stress disorder (PTSD) or clinically relevant posttraumatic stress symptoms (PTSS) in preschoolers with injuries following accidental trauma, such as road traffic or burn accidents. In consequence, secondary preventive efforts (early interventions) should be undertaken to minimize such long-term deleterious consequences in children. While important components of successful early interventions have been identified in school-age children, evidence is completely lacking for younger children, especially for those below the age of 4 years.

Aims: The proposed study aims at examining the effect of a newly developed, standardized early psychological intervention in reducing posttraumatic maladjustment and in enhancing health-related quality of life in children ages 1 to 4 years with acute burn injuries. Also, the effectiveness of an early screening measure in identyfing children with high risk for psychological follow-up problems shall be studied.

Method: The study is designed as a randomized controlled trial within a stepped procedure. First, eligible children will be screened 5 to 7 days post injury by means of a standardized measure for their risk of developing PTSS. After a baseline assessment, children at risk will then be randomly allocated to either a control group (standard medical care) or an intervention group. Participants of the intervention group will be provided with the standardized "EPICAP 1-4" intervention which uses established cognitive-behavioral techniques and is directed to the parents. The intervention includes the following components: psychoeducation on child and parental PTSS, promotion of adaptive strategies to manage child and parental distress, construction of a parental trauma narrative, promotion of strategies that increase parental capacity and enhance parent-child relationship. The intervention consists of two face-to-face sessions with the parents (at baseline and 1 week later) and a follow-up call or short follow-up face-to-face meeting (6 weeks after the first session). Blinded follow- up assessments with standardized parent report measures will be conducted at 3 and 6 months post injury. The primary outcome measures are child PTSD and PTSS, secondary outcome measures include child behavior and health-related quality of life. In addition, a variety of socio-demographic, medical and parental variables will be assessed as co-variates. Children screened as low-risk will be reassessed only at 6 months to make sure that the screening procedure is valid.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1- 4 years
* Acute burn injury
* Treatment at University Children's Hospital Zurich

Exclusion Criteria:

* severe comorbid head injury in the child (Glasgow Coma Scale < 9)
* expected initial stay in the pediatric intensive care unit for more than a week
* burn injury due to suspected or substantiated child abuse
* any previous evidence of cognitive impairment or pervasive developmental disorder in the child
* insufficient command of the German language in both parents

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
DIPA PTSD Module | 6 months
  The DIPA PTSD module is an interview of caregivers for children from nine months to six years old that assesses DSM-5 PTSD preschool criteria.

SECONDARY OUTCOMES:
Child Behavior Checklist 11⁄2-5 (CBCL; Achenbach & Rescorla, 2000) | 6 months
  This is a highly standardized, widely used and well validated 100-item parent-report measure for children ages 1.5 to 5 years.3 Caregivers have to report the extent to which they agree with statements on a 3-point Likert scale ranging from 1 (not true) to 3 (very true). The questionnaire yields scores for two broad-band sca- les (internalizing and externalizing behavior problems), and an overall total behavioral problems score.
TNO-AZL Preschool Children Quality of Life Questionnaire (TAPQOL; Fekkes et al., 2000). | 6 months
  The TAPQOL is a 43-item multidimensional instrument that yields sum scores for physical, emotional, social, and cognitive functioning by parent report. Also, an overall sum score indicating general HRQoL can be computed. The TAPQOL can be applied to children of 9 months to 6 years of age. It has good construct, criterion, and concurrent validity and a good internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Markus A. Landolt, PhD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haag AC, Landolt MA. Young Children's Acute Stress After a Burn Injury: Disentangling the Role of Injury Severity and Parental Acute Stress. J Pediatr Psychol. 2017 Sep 1;42(8):861-870. doi: 10.1093/jpepsy/jsx059. PMID 28340168
- [Background] De Young AC, Haag AC, Kenardy JA, Kimble RM, Landolt MA. Coping with Accident Reactions (CARE) early intervention programme for preventing traumatic stress reactions in young injured children: study protocol for two randomised controlled trials. Trials. 2016 Jul 28;17:362. doi: 10.1186/s13063-016-1490-2. PMID 27464735
- [Derived] Haag AC, Landolt MA, Kenardy JA, Schiestl CM, Kimble RM, De Young AC. Preventive intervention for trauma reactions in young injured children: results of a multi-site randomised controlled trial. J Child Psychol Psychiatry. 2020 Sep;61(9):988-997. doi: 10.1111/jcpp.13193. Epub 2020 Jan 8. PMID 31912485